CLINICAL TRIAL: NCT00798512
Title: DESERVE: Diffusion Weighted-MRI Based Evaluation of the Effectiveness of Endovascular Clamping During Carotid Artery Stenting With the Mo.Ma Device. A Prospective, Multicenter Study.
Brief Title: Diffusion Weighted-MRI Based Evaluation of the Effectiveness of Endovascular Clamping During Carotid Artery Stenting With the Mo.Ma Device.
Acronym: DESERVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Invatec S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: N999
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Carotid Artery Disease; Stroke Prevention
Keywords: carotid artery stenting; cerebral protection; stroke; ischemic lesion; DW-MRI
MeSH Terms: conditions — Carotid Artery Diseases; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Single arm Study in which 120 patients fulfilling eligibility criteria will be screened and undergo carotid stenting with the Cristallo ideale™ carotid stent after placement of the Mo.Ma device as cerebral protection system. The technique of diffusion-weighted magnetic resonance imaging (DW-MRI) will be used to identify new ischemic lesions.
  Interventions: Device: Carotid artery stenting

INTERVENTIONS:
Device: Carotid artery stenting — The MO.MA is a cerebral protection catheter based on the proximal flow blockage concept which is achieved by endovascular clamping of Common Carotid Artery (CCA) and External Carotid Artery (ECA). The MO.MA proximal flow blockage cerebral protection device is indicated to be used in patients eligible for carotid angioplasty and/or the carotid bifurcation and is aimed to prevent brain embolism during the stenting procedure.
  For the purpose of this study the Cristallo Ideale™ Carotid Stent System (Invatec S.R.L. Roncadelle, Italy) will be exclusively used. Cristallo Ideale™ consists of a carotid dedicated self-expanding stent pre-mounted on a rapid exchange delivery catheter. The stent platform is made of a Nitinol alloy and characterized by a hybrid design with closed cell in the central zone and open cell in both end zones (proximal and distal).

SUMMARY:
The purpose of this study is to detect new ischemic lesions after carotid artery stenting (with the Cristallo Ideale stent), in patients with high grade carotid artery stenosis, by diffusion-weighted magnetic resonance imaging (DW-MRI), using the endovascular proximal flow blockage (Mo.Ma device) for cerebral protection.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old;
2. Eligibility for carotid artery revascularization;
3. A significant stenosis in symptomatic patients with ≥ 50% Diameter Stenosis (%DS) or asymptomatic ≥ 80 %DS as defined by angiography.

   Symptomatic is defined as a carotid artery stenosis associated with ipsilateral TIA, amaurosis fugax, ischemic stroke or retinal infarction within 6 months prior to enrollment.
4. Suitable clinical conditions to perform DW-MRI.
5. Written informed consent as approved by the Ethics Committee of the respective clinical site.

Exclusion Criteria:

1. Female with childbearing potential without a negative pregnancy test.
2. Life-expectancy less than 6 months.
3. Underlying disease of the carotid artery other than atherosclerosis (e.g. vasculitis, traumatic dissection, fibromuscular dysplasia).
4. Prior stenting in the target vessel;
5. Patients with chronic or re-current atrial fibrillation.
6. Patient has had a Myocardial Infarction within 72 hours prior to the procedure.
7. Patient experienced a stroke within 4 weeks prior to the procedure.
8. History of severe disabling stroke according to the modified Rankin scale > 4.
9. Severe renal failure (serum creatinine > 2.0 mg/dL).
10. Severe peripheral arterial occlusive disease, which might impede a safe introduction of a 9F-sheath for the use of a Mo.Ma-device.
11. Any known allergies and / or intolerances to the following: ASA, Clopidogrel, Statins, Heparin, Nitinol, contrast agents (that cannot be adequately pre-medicated).
12. Patient currently participating in an investigational drug or device study which has not reached the primary endpoint yet or which clinically interferes with the DESERVE study endpoints.
13. Any planned major surgery within 30 days after the study procedure.
14. In the investigators opinion patient has a severe co-morbid condition(s) that could limit the ability to participate in the study.

    Angiographic exclusion criteria:
15. Totally occluded internal carotid artery considered as the target vessel.
16. Multiple internal carotid artery stenoses or lesion longer than 4 cm (whichever occurs) that cannot be covered by one (1) stent.
17. Severe ostial stenosis of the common carotid artery.
18. The presence of ipsilateral intracranial stenosis that requires treatment.
19. Contralateral occlusion of the internal carotid arteries associated with a poor collateral flow through the circle of Willis.
20. An aortic arch anatomical complexity that may preclude the safe placement of the Mo.Ma device including particularly, the impossibility to navigate a stiff guide wire into the external carotid artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The de-novo occurrence of intra-cerebral lesions per patient by comparing baseline (within 1 week prior procedure) and post-procedural DW-MRI (from 3 to 12 hours post procedure). | 3-12 hours after index procedure

SECONDARY OUTCOMES:
Device Success; Technical Success; Procedural Success; Restenosis rate at 30 days follow up; TLR at 30 days follow up; Access Site Complications; MACCE at 30 days; Incidence of TIA up to 30 days. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Biamino, MD, Study Chair — Gruppo Villa Maria - Endovascular Villa Maria Cecilia Hospital
Locations (6):
- Germany (2):
  - CardioVascular Center Frankfurt, Sankt Katharinen, Frankfurt
  - Heart Center Leipzig, Clinical and Interventional Angiology, Leipzig
- Italy (3):
  - Casa di Cura Privata "Montevergine" S.p.A., Mercogliano, Avellino
  - Gruppo Villa Maria, Villa Maria Cecilia Hospital, Cotignola, RA
  - Ospedale Civile di Mirano, Unità di Cardiologia, Mirano
- Jagellonian University, College of Medicine, Institute of Cardiology, University Hospital, Krakow, Poland